CLINICAL TRIAL: NCT05554627
Title: VA Aripiprazole vs. Esketamine for Treatment of Depression VAST-D II
Brief Title: VA Aripiprazole vs Esketamine for Treatment Resistant Depression
Acronym: VAST-D II
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study funding was withdrawn by study sponsor (CSR&D) prior to enrollment due to budget constraints.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEP-002-20S
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Esketamine; Ketamine; Aripiprazole; aripiprazole lauroxil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study will be open-label where both the treating staff and the participant are unblinded to their treatment assignment, but the primary outcome will be assessed via telehealth by blinded remote raters without knowledge of treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esketamine (Experimental): Intranasal spray of esketamine. Administered twice weekly for first 4 weeks, reduced to once weekly until week 12, then dosage will be determined by response and treating prescriber.
  Interventions: Drug: Esketamine
- Aripiprazole (Active Comparator): Participants will be randomized in a 1:1 ratio of equal allocation to either adjunctive ARI (n=470) or adjunctive IN ESK (n=470), stratified by participating site.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Esketamine — Intranasal spray; a dissociative hallucinogen drug used as a general anesthetic and an antidepressant for treatment of depression.
  Other Names: Spravato (for depression), Ketanest (for anesthesia)
  Arms: Esketamine
Drug: Aripiprazole — Atypical antipsychotic; used in the treatment of schizophrenia and bipolar disorder. Other uses include as an add-on treatment in major depressive disorder, tic disorders and irritability associated with autism. Taken by mouth or injection into a muscle.
  Other Names: Abilify, Aristada
  Arms: Aripiprazole

SUMMARY:
This is an open-label, parallel-group, randomized clinical trial of up to 6 months treatment of adjunctive intranasal (IN) esketamine (ESK) vs. adjunctive aripiprazole (ARI) in Veterans with unipolar Treatment Resistant Depression (TRD). This study will assess the efficacy, safety, and acceptability of adjunctive IN ESK in comparison to ARI, one of the best studied and most widely used adjunctive therapies for TRD. The primary hypothesis is that participants receiving adjunctive IN ESK will be significantly more likely to achieve remission after six weeks of treatment as compared to those who receive adjunctive ARI. Depressive symptoms will be assessed by central raters (CR), blinded to treatment assignment, using the clinician rated version of the Quick Inventory of Depressive Symptomatology (QIDS-C16), a well-validated tool that is commonly used and is easily translated across other depression inventory scales. The study is powered to detect an absolute difference in remission rates of 10%, or larger, at 6 weeks. Additional outcomes of interest include symptom reduction across 6 months of randomized therapy, side effects and other tolerability indices, attrition rates and measures of quality of life and cost-effectiveness.

DETAILED DESCRIPTION:
OVERVIEW: This is an open-label, parallel-group, randomized clinical trial of up to 6 months treatment of adjunctive intranasal (IN) esketamine (ESK) vs. adjunctive aripiprazole (ARI) in Veterans with unipolar Treatment Resistant Depression (TRD). This study will assess the efficacy, safety, and acceptability of adjunctive IN ESK in comparison to ARI, one of the best studied and most widely used adjunctive therapies for TRD. The primary hypothesis is that participants receiving adjunctive IN ESK will be significantly more likely to achieve remission after six weeks of treatment as compared to those who receive adjunctive ARI. Depressive symptoms will be assessed by central raters (CR), blinded to treatment assignment, using the clinician rated version of the Quick Inventory of Depressive Symptomatology (QIDS-C16), a well-validated tool that is commonly used and is easily translated across other depression inventory scales. The study is powered to detect an absolute difference in remission rates of 10%, or larger, at 6 weeks. Additional outcomes of interest include symptom reduction across 6 months of randomized therapy, side effects and other tolerability indices, attrition rates and measures of quality of life and cost-effectiveness.

BACKGROUND: Among all medical, mental health and substance related disorders, Major Depressive Disorder (MDD) is a leading cause of disease burden worldwide. MDD is a major cause of suffering and disability for those receiving their care from the Veterans Health Administration (VHA). Depression not only can have a ruinous effect on quality of life and economic productivity, but also adversely effects health and reduces lifespan by 10 years. About 2/3rds of those who die by suicide have a depressive disorder. The best means to reduce the disease burden associated with MDD centers around prompt recognition and vigorous pharmacologic and/or psychotherapeutic treatment. Many reasonably safe antidepressants and effective forms of psychotherapy are available, but about one-third of depressed patients do not respond to these therapies. By regulatory convention, the term TRD is used when a depressed patient has not responded to two or more adequate medication trials in the current episode. So defined, patients with TRD account for a disproportionately large share of treatment resources and, despite such efforts, are at the highest risk to become chronically ill, develop a complicating substance abuse disorder and/or die by suicide. In response to the urgent need to test promising approaches to improve the outcomes of depressed Veterans, in 2010 the VA Cooperative Studies Program initiated the VA Augmentation and Switching Treatments for Improving Depression Outcomes (VAST-D) study. Focusing on the most promising strategies available at the time, VAST-D enrolled 1,522 patients who had failed to respond to their previous antidepressant treatment. Participants were randomized to one of three strategies: adjunctive ARI, switching from their current antidepressant to bupropion or adding adjunctive bupropion. The results of VAST-D, published in JAMA in August 2017, showed that adjunctive ARI resulted in a significantly greater likelihood of remission as compared to switching to bupropion; the group receiving adjunctive bupropion tended to have intermediate outcomes. Secondary analyses of VAST-D demonstrated that the advantage of adjunctive ARI among 12-week remitters was sustained across up to six months of therapy and was evident whether or not patients had co-occurring PTSD. The critical importance of VAST-D is that it was the first study to show any distinct advantage for any "next step" treatment of MDD over any other and thus raised the hope that additional improvements could be found.

Separately, a series of studies showed that intravenous infusions of the dissociative anesthetic ketamine could produce rapid antidepressant effects in a meaningful subset of patients with TRD. Many patients begin to respond to infusions of sub-anesthetic doses of racemic ketamine (i.e., 0.5 mg/kg) within 24 hours of administration and, although the effects have been transient, most patients experience 4-7 days of symptom relief with each infusion. Although such off-label use of this Schedule III controlled substance has increased in the past decade, it is still rarely used, and issues pertaining to the feasibility of an infusion therapy in ambulatory psychiatric care settings and abiding concerns about the lack of well-controlled efficacy and safety data pertaining to longer term use have not been addressed. Most recently, the efficacy and safety of IN delivery of the "s" enantiomer of racemic ketamine (a.k.a. 'esketamine' [ESK]) has been evaluated as a means to address these concerns. The safety and efficacy of ESK was evaluated in a series of phase III studies that ultimately led to the recent approval by the U.S. FDA of ESK (Spravato) for the treatment of TRD in adults. The FDA evaluated ESK in the context of three 4-week, placebo-controlled, parallel-group studies (Studies 3001 and 3002 in adults 18 to 65 years of age; Study 3005 in patients 65 years or older) and one longer-term randomized withdrawal study (Study 3003). Long-term safety was also evaluated in a 12-month open-label safety study (Study 3004). In aggregate, the FDA determined that the available evidence provided substantial evidence of efficacy together with an acceptable risk profile. Despite this important potential advance in the treatment of depression, no study has evaluated the efficacy and safety of esketamine in a VA population. No study has evaluated ESK in comparison to an alternative pharmacotherapy for TRD, and no study has systematically examined outcomes and adverse effects for up to 6 months, a critical need in a chronic illness.

OBJECTIVE: The aim of VAST-D II is to study the efficacy and safety of adjunctive IN ESK as a treatment option for patients with TRD. Specifically, this study is designed to assess the efficacy of adjunctive IN ESK, in comparison to the best validated "next step" pharmacotherapy for Veterans with TRD, namely adjunctive oral ARI. The primary outcome is remission in a short-term acute treatment phase of six weeks. The key secondary outcome is reduction in depressive symptoms from baseline to long-term follow-up of six months. The extended follow-up period is also essential to collect important data on the effectiveness, safety, and acceptability of this novel treatment in the investigators' patient population. Exploratory outcomes include comparisons of symptom improvement, remission rates, and relapse rates after remission, PTSD symptoms, suicidality, quality of life, and cost-benefit analysis.

RESEARCH PLAN: 940 participants will be recruited from approximately 25 VA medical centers, over an estimated 38 months, with each participant being treated and followed for 6 months. All participants will be screened for eligibility including MDD diagnosis, TRD defined as at least two unsuccessful trials on a pharmacological antidepressant, suicidal ideation (SI) levels, current levels of substance abuse, and stability of medical condition. Otherwise, the eligibility criteria are posed with an interest in capturing a largely representative sample.

Participants will be randomized in a 1:1 ratio of equal allocation to either adjunctive ARI (n=470) or adjunctive IN ESK (n=470), stratified by participating site. This study will be open-label where both the treating staff and the participant are unblinded to their treatment assignment, but the primary outcome will be assessed via telehealth by blinded remote raters without knowledge of treatment assignment. All participants will complete in person or telehealth follow-ups at weeks 1, 2, 3, 4, 6, 8, 10, 12, 18, and 24. The primary outcome will be remission at week 6 defined by a QIDS-C16 score 5 assessed by blinded-to-treatment raters remotely by telehealth.

Based on the week 6 findings of VAST-D, the investigators anticipate that about 16% of TRD patients will remit with adjunctive ARI. The investigators predict that a 6-week course of adjunctive IN ESK will result in at least a 26% remission rate. A total sample size of 940 participants will be required to test the hypothesis of a 10% absolute difference in proportions at 90% power given a two-sided type-I error =0.05, adjusting for crossovers and losses (25%).

IMPACT: A major comparative efficacy study of adjunctive IN ESK vs. the next best strategy, adjunctive ARI, in Veterans with TRD is urgently needed to identify the short and longer-term benefits and risks of esketamine, and whether the overall gains are substantial enough to offset side effects, drug and treatment-associated costs, and patient burden incurred by the need for ESK dosing in a healthcare setting and subsequent on-site monitoring.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of current episode of major depressive disorder (MDE, single or recurrent, non-psychotic) by MINI
* TRD defined as at least 2 failed trials of antidepressants (adequate dose and duration) including the current episode and another during last 2 years
* Current QIDS-C16 score of > 14
* Currently on an antidepressant medication at stable dose for at least 6 weeks without adequate improvement
* Ages 18-74 years old at the time of randomization

Exclusion Criteria:

* Lifetime history of bipolar disorder, schizophrenia, schizoaffective disorder, or other psychotic disorder
* Presence of psychotic features in the current MDE
* Lifetime history of major neurocognitive disorder or any diagnosed neurodegenerative or neurodevelopmental disorder
* Current evidence of cognitive dysfunction based on MoCA score < 24
* Hypersensitivity to ESK or ketamine
* History of aneurysmal vascular disease or arteriovenous malformation
* History of intracerebral hemorrhage
* Uncontrolled hypertension (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg, unless cleared by the patient's primary care physician)
* History of significant cardiovascular disease, including recent myocardial infarction (within last 12 months), unstable angina, or chronic heart failure
* History of interstitial or ulcerative cystitis
* Any current unstable medical condition that in the opinion of the investigator would place the patient at increased risk, including hepatic, respiratory, immunological, cardiovascular, endocrine, or renal disease
* Imminent need for psychiatric hospitalization
* History of moderate or severe SUD in last 6 months will be excluded, not including cannabis, tobacco, and caffeine
* Women who are pregnant, lactating, or planning to become pregnant or those of childbearing potential who are sexually active but unwilling to use a contraceptive
* Unable to provide informed consent
* Current treatment with any antipsychotic
* Prior antidepressant treatment with ketamine or ESK within the current episode/past two years
* Prior antidepressant treatment with ARI at an FDA-approved dose for at least 6 weeks within the past 2 years
* Lifetime history of ketamine use disorder
* History of drug induced leukopenia

For women of childbearing potential, pregnancy will be excluded prior to randomization and counseling on potential risks of taking ESK or ARI during pregnancy will be provided.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptoms (QUIDS-C16) | 6 Weeks
  Scale of depressive symptoms at six weeks post-randomization. QUIDS is the 16-item Quick Inventory of Depressive Symptomology. Total QUIDS scores range from 0 to 27. Higher values indicate worse depression symptoms/worse outcome. Scores of 5 or lower are indicative of no depression; scores from 6 to 10 are indicative of mild depression; 11 to 15 indicate moderate depression; 16 to 20 reflects severe depression, and total scores greater than 21 indicate very severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Somaia Mohamed, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (26):
- United States (26):
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - CERC (VISN1, West Haven, CT), West Haven, Connecticut
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Jackson C. Montgomery VA Medical Center, Muskogee, OK, Muskogee, Oklahoma
  - Philadelphia MultiService Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - Salem VA Medical Center, Salem, VA, Salem, Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No